CLINICAL TRIAL: NCT01826994
Title: Incremental Value of Heart-type Fatty Acid-Binding Protein (H-FABP) in Evaluating Patients Presenting With Symptoms Possibly Matching Acute Coronary Syndrome in Primary Care
Brief Title: Incremental Value of Point of Care H-FABP Testing in Primary Care Patients Suspected of Acute Coronary Syndrome
Acronym: RAPIDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: FABPulous B.V. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-3-015; ABR registry (Registry Identifier: ABR registration NL43078.068.12)
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Acute Coronary Syndrome; Angina Pectoris, Unstable; Angina Pectoris, Stable; Thoracic Diseases
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Angina, Stable; Thoracic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients (Other): heart type fatty acid binding protein testing
  Interventions: Device: heart type fatty acid binding protein testing

INTERVENTIONS:
Device: heart type fatty acid binding protein testing

SUMMARY:
Rationale:

Thoracic complaints, possibly due to a cardiac ischemic cause are a diagnostic challenge in general practice. When an underlying ischemic cardiac condition (AMI (acute myocardial infarction), UAP (unstable angina pectoris)) is considered, referral from general practitioner (GP) to a cardiologist has to take place. However, cardiac analysis in 80% of referred patients is negative. To optimize referral decisions of GPs, new and fast diagnostics are needed.

Objective:

To assess the incremental diagnostic value for AMI of a novel rapid PoC H-FABP-test in addition to history taking and physical examination in patients presenting in daily general practice with possible AMI. In addition the cost-effectiveness of the test will be evaluated.

Study design:

Delayed type cross-sectional diagnostic study.

Study population:

Patients presenting to the GP with any new-onset chest complaint, at time of presentation not lasting for more than 24 hours, that is considered to be of possible cardiac origin by the GP.

Intervention:

Point of care Heart Type Fatty Acid Binding Protein test (PoC H-FABP-test), added to usual care. PoC H-FABP-testing, by qualitatively measuring H-FABP in one single drop of blood obtained by finger prick, is added to normal procedures of consultation and referral decision by the GP.

Main study parameters / endpoints:

Sensitivity, specificity, positive and negative predictive value of point of care H-FABP-testing for AMI, alone as well as part of a clinical diagnostic algorithm, in patients with thoracic complaints in general practice. All outcome measures, based on using an algorithm and/or point of care H-FABP-testing, will be compared to regular diagnostic assessment by the GP without using an algorithm and/or point of care H-FABP-testing. Therefore, incremental value of H-FABP-testing and/or a diagnostic algorithm is measured.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Individual participants will experience low risk, since study participation comprehends regular care except for an extra finger prick and possibly collection of one extra venous blood sample. For this low amount of disadvantage, the participant will experience no advantage either. However, results of the study will possibly be useful for similar patients in future.

ELIGIBILITY:
Inclusion Criteria:

* new-onset chest complaint, considered to be of possible cardiac origin by the general practitioner
* In case of death of identified cause patients are included as well.

Exclusion Criteria:

* all attention has to be on acute support for the patient
* symptoms are present for more than 24 hours
* oral informed consent is not given during presentation
* written informed consent is refused afterwards
* a traumatic cause is present
* complaints are presented that can be regarded as a recurrence of earlier complaints with clear diagnosis in the past
* death of unidentified cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
diagnostic value of point of care heart type fatty acid binding protein testing for acute myocardial infection, alone as well as in combination with a clinical diagnostic algorithm | one and a half year
  Sensitivity, specificity, positive and negative predictive value of point of care heart type fatty acid binding protein testing for acute myocardial infection, alone as well as in combination with a clinical diagnostic algorithm. To determine influence of sex, age, duration of the complaints, and kidney function on clinical performance of heart type fatty acid binding protein testing, subgroup analysis within our study population will be performed

SECONDARY OUTCOMES:
cost-effectiveness | one and a half year
  An economic evaluation by means of an incremental cost-effectiveness ratio will be performed. This evaluation will be performed by determination of the ratio between the difference in costs and the difference in benefits between the two strategies that are observed in this study, being the usual reference policy of the general practitioner and the reference policy that could be created when a determined algorithm combined with point of care heart type fatty acid binding protein testing would be used.
definition of an algorithm towards diagnosing acute coronary syndrome and unstable angina | one and a half year
  Predictive value of a diagnostic algorithm towards diagnosing acute coronary syndrome and unstable angina is determined, since unstable angina is a condition without rise in biomarkers, but should not be missed by a general practitioner assessing thoracic complaints

CONTACTS AND LOCATIONS:
Overall Officials: Geert Jan Dinant, professor, Study Chair — Maastricht University
Locations (7):
- ACHG, Leuven, Vlaams Brabant, Belgium
- Netherlands (6):
  - HOZL, Heerlen, Limburg
  - ZIO, Maastricht, Limburg
  - Omnes, Sittard, Limburg
  - Cohesie, Venlo, Limburg
  - BeRoEmD, 's-Hertogenbosch, North Brabant
  - SGE, Eindhoven, North Brabant

REFERENCES:
- [Derived] Willemsen RT, Buntinx F, Winkens B, Glatz JF, Dinant GJ; 'RAPIDA'-study team. The value of signs, symptoms and plasma heart-type fatty acid-binding protein (H-FABP) in evaluating patients presenting with symptoms possibly matching acute coronary syndrome: background and methods of a diagnostic study in primary care. BMC Fam Pract. 2014 Dec 12;15:203. doi: 10.1186/s12875-014-0203-8. PMID 25738970